CLINICAL TRIAL: NCT04282915
Title: Reducing Stigma Among Healthcare Providers to Improve Mental Health Services: Cluster Randomized Controlled Trial (RESHAPE-cRCT)
Brief Title: Reducing Stigma Among Healthcare Providers (RESHAPE-cRCT)
Acronym: RESHAPE-cRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Duke University (Other); Transcultural Psychosocial Organization Nepal (Other); King's College London (Other)
Responsible Party: Principal Investigator, Brandon A Kohrt, MD, PhD, Associate Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: R01MH120649 (NIH)
Record Dates: First submitted 2020-02-19; First posted 2020-02-25 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Mental Disorder; Depressive Disorder; Anxiety Disorder; Alcohol Use Disorder; Psychotic Disorders
Keywords: Primary care; Stigma; Developing countries; Mental health
MeSH Terms: conditions — Mental Disorders; Depressive Disorder; Anxiety Disorders; Alcoholism; Psychotic Disorders; Social Stigma; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized controlled trial with municipalities being the unit of randomization. 24 municipalities will be randomized to either RESHAPE or implementation as usual. Three health facilities in each municipality will participate in the study. All primary care providers with prescribing rights will be trained based on their municipality randomization arm.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: There are two types of study participants: primary care providers and primary care patients. Based on the municipality of randomization, primary care providers will either participate in RESHAPE training or implementation as usual training. Patients will not be randomized because the health facilities they attend are already assigned to either having the primary care providers trained through RESHAPE or implementation as usual. The providers and patients will be masked to the implementation, i.e., they will not be given information on the differences in the two different implementation strategies. Research assistants and research psychiatrists who conduct the assessments will be masked to whether the provider or patients are in the RESHAPE or implementation-as-usual arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation as Usual (Active Comparator): Primary care providers will be trained in the 7-day curriculum of the mental health Gap Action Programme adapted by the Nepal Ministry of Health.
  Interventions: Other: mental health Gap Action Programme
- RESHAPE (Experimental): Primary care providers will be trained in the 7-day curriculum of the mental health Gap Action Programme, plus they will have co-facilitation by mental health service users providing recovery testimonials as well as aspirational figures presenting testimonies and conducting myth-busting sessions.
  Interventions: Other: Reducing Stigma among Healthcare Providers (RESHAPE); Other: mental health Gap Action Programme

INTERVENTIONS:
Other: Reducing Stigma among Healthcare Providers (RESHAPE) — Mental health service users are trained using Photo Voice to develop recovery story testimonials. They then participate in primary care providers mental health Gap Action Programme training. In addition, aspirational figures are trained to provider testimonials and conduct myth-busting.
  Arms: RESHAPE
Other: mental health Gap Action Programme — The mental health Gap Action Programme is a training program for primary care providers in mental health services. The curriculum has been developed by the World Health Organization and was adapted in Nepal and certified by the Ministry of Health.

SUMMARY:
A growing number of trials have demonstrated treatment effectiveness for mental illness by non-specialist providers, such as primary care providers, in low-resource settings. A barrier to scaling up these evidence-based practices is the limited uptake from trainings into service provision and lack of fidelity to evidence-based practices among non-specialists. This arises, in part, from stigma among non-specialists against people with mental illness. Therefore, interventions are needed to address attitudes among non- specialists. To address this gap, REducing Stigma among HeAlthcare Providers to improvE Mental Health services (RESHAPE), is an intervention for non-specialists in which social contact with persons with mental illness is added to training and supervision programs. A cluster randomized control trial will address primary objectives including changes in stigma (Social Distance Scale) and improved quality of mental health services, operationalized as accuracy of identifying patients with mental illness in primary care. The control condition is existing mental health training and supervision for non-specialists delivered through the Nepal Ministry of Health's adaptation of the World Health Organization mental health Gap Action Programme. The intervention condition will incorporate social contact with people with mental illness into existing training and supervision. Participants in the cluster randomized control trial will be the direct beneficiaries of training and supervision (primary care providers) and indirect beneficiaries (their patients). Primary care workers' outcomes include stigma (Social Distance Scale), knowledge (mental health Gap Action Programme knowledge scale), implicit attitudes (Implicit Association Test), clinical self-efficacy (mental health Gap Action Programme knowledge scale), and clinical competence (Enhancing Assessment of Common Therapeutic factors) to be assessed pre-training, post-training, and at 3- and 6-month follow-up. Accuracy of diagnoses will be determined through the Structured Clinical Interview for the Diagnostic and Statistical Manual version 5, which will be assessed at 3 months after patient enrollment. Patient outcomes include functioning, quality of life, psychiatric symptoms, medication side effects, barriers to care, and cost of care assessed at enrollment and 3 and 6 months. This study will inform decisions regarding inclusion of persons living with mental illness in training primary care providers.

DETAILED DESCRIPTION:
There continues to be a major gap between the global burden of persons with mental illness and the number of patients receiving adequate treatment. In the U.S. and other high-income countries, approximately 1 out of 5 persons receives minimally adequate care. In lower-middle income countries, it ranges from 1 out of 27 to 1 out of 100 persons. To address this gap in low- and middle-income countries, a key strategy has been the use of primary care health workers to detect and deliver of care for mental illness. The World Health Organization has developed the mental health Gap Action Programme to train primary care workers to detect mental illness and deliver evidence-supported treatment. However, research to date suggests that implementation strategies for mental health Gap Action Programme are inadequate as evidenced by low detection rates. In Nepal, fewer than half of persons with mental illness were correctly identified by mental health Gap Action Programme-trained primary care workers. A potential barrier to effective implementation of primary care detection is stigma among primary care workers against persons with mental illness.

Our preliminary work suggests that reducing primary care workers' stigma against persons with mental illness may improve accurate detection of mental illness. A version of the mental health Gap Action Programme training that includes a stigma reduction component was developed: REducing Stigma among HealthcAre ProvidErs (RESHAPE). In RESHAPE, persons with mental illness (i.e., service users) are trained to share recovery stories, conduct myth-busting sessions, and promote mental health advocacy. A pilot cluster randomized controlled trial was conducted in Nepal comparing standard mental health Gap Action Programme training delivered psychiatrists and psychosocial specialists with a mental health Gap Action Programme training delivered by both specialists and service users (RESHAPE). Consistent with high-income country literature demonstrating that interaction with service users reduces stigma more effectively that only providing knowledge, stigma was lower among the RESHAPE- arm trained health workers. The pilot results also suggest that reducing stigma may improve detection of mental illness. Therefore, involvement of mental health service users in training primary care workers may reduce stigma, and that stigma reduction may mediate improved detection of mental illness. If these findings are confirmed in an appropriately powered cluster randomized controlled trial, this service user collaborative implementation strategy could make a major contribution to improving primary care detection in low- and middle-income countries, as well as in the U.S. A hybrid implementation-effectiveness (type-3) cluster randomized controlled trial will be in Nepal comparing mental health Gap Action Programme standard implementation with the RESHAPE implementation strategy. Our team of U.S. and Nepali researchers, in partnership with the Nepal Ministry of Health, demonstrated the feasibility of the cluster randomized controlled trial design and identified strategies for cost effectiveness modeling. Target conditions will be depressive disorder, psychotic disorders, and alcohol use disorder.

Aim 1 - To evaluate the impact of the RESHAPE service user engagement on stigma among primary care workers. Hypothesis: Primary care workers in the RESHAPE arm will have less stigma toward persons with mental illness (measured with the Social Distance Scale) 3 months after training compared with primary care workers in the standard training.

Aim 2 - To evaluate the impact of the RESHAPE training on accuracy (sensitivity and specificity) of detection, as measured by the proportion of true positive and true negative diagnoses among patients presenting to primary care facilities, as confirmed by a psychiatrist's structured clinical interview; and to evaluate stigma as a mediator of differences in accuracy. Hypothesis: Primary care workers in the RESHAPE arm will have greater accuracy of detecting mental illness. Secondary analyses: implementation arm differences in patient quality adjusted life years and cost utility will be evaluated.

ELIGIBILITY:
**Primary Care Providers**

Inclusion Criteria:

* All health workers from the facilities included in the study will be invited to participate
* Health workers will be between 18 and 65 years of age based on employment criteria
* within the government health system.
* All participants will need to have Nepali language competency,
* be actively engaged in care provision in their health cluster,
* have a valid certificate of practice from the Ministry of Health
* Health workers will need to have permission from their health supervisor to attend the entire duration of the training,

Exclusion Criteria:

* any prior citations on their clinical practice licensure or any other government credentialing violations.

**Patients**

Inclusion Criteria:

* All patients (with non-emergency medical needs) presenting to the primary care
* any of the following groups:
* (a) any mental illness diagnosis including depression, psychosis (bipolar disorder with a manic episode, schizophrenia, major depressive disorder with psychotic features, and alcohol use disorder with psychosis) and alcohol use disorder; plus the other conditions included in Nepal's mental health Gap Action Programme: anxiety, conversion, epilepsy, dementia, child and adolescent, other substance abuse (these patients are included because misdiagnosis is common with regard to missing or overdiagnosing one condition in place of another mental illness); comorbid conditions are also acceptable;
* (b) any patients screening above cut-off scores on the tools; and
* (c) 10% of patients who are negative on all of the above criteria.
* any patients previously treated for mental illness would be included
* age range will be 16 years or older, with no upper age limit (mental health Gap Action Programme training covers child and adolescent through mental illnesses affecting elderly population).
* all participants will be able to speak Nepali
* able to complete the research interview with the research assistants who will read all of the assessment tools.

Exclusion Criteria:

* Patients with immediate medical needs requiring referral and emergency services (e.g., serious injury; pre-eclampsia; dehydration; status epilepticus)
* patients needing acute psychiatric services (e.g., suicide attempts, alcohol withdrawal, psychosis/mania that cannot be managed in a community setting) who are referred for immediate hospitalization
* Patients under the age of 16 years old will be excluded

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8705 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Social Distance Scale (SDS) | 6 months post training
  12-item scale of willingness to interact with persons with mental illness, minimum = 0, maximum = 72, higher score is worse outcome
Structured Clinical Interview for Diagnostic and Statistical Manual 5 (SCID-5) | 3-months post-patient enrollment
  Accuracy of clinical decision making (this a diagnostic tool, there are no maximum or minimum scores, the objective is to determine if an appropriate diagnosis is selected that will lead to appropriate management)

SECONDARY OUTCOMES:
mental health Gap Action Programme knowledge test | 6 months post-training
  Multiple-choice assessment from mental health Gap Action Programme training materials; minimum = 0, maximum = 100, higher is better outcome
mental health Gap Action Programme knowledge test | 3 months post-training
  Multiple-choice assessment from mental health Gap Action Programme training materials, minimum = 0, maximum = 100, higher is better outcome
mental health Gap Action Programme knowledge test | immediately after the training
  Multiple-choice assessment from mental health Gap Action Programme training materials, minimum = 0, maximum = 100, higher is better outcome
mental health Gap Action Programme self-efficacy assessment | 6-months post-training
  Self-reported clinical efficacy for mental health services, minimum = 0; maximum = 5, higher score is better outcome
mental health Gap Action Programme self-efficacy assessment | 3-months post-training
  Self-reported clinical efficacy for mental health services, minimum = 0; maximum = 5, higher score is better outcome
mental health Gap Action Programme self-efficacy assessment | immediately after the training
  Self-reported clinical efficacy for mental health services, minimum = 0; maximum = 5, higher score is better outcome
Implicit Association Test | 6-months post-training
  Computer-based neuropsychological assessment of implicit bias related to mental illness, there is no maximum or minimum score, score is D-score based on comparison of timing; positive scores equal more bias
Implicit Association Test | 3-months post-training
  Computer-based neuropsychological assessment of implicit bias related to mental illness, there is no maximum or minimum score, score is D-score based on comparison of timing; positive scores equal more bias
Implicit Association Test | immediately after the training
  Computer-based neuropsychological assessment of implicit bias related to mental illness, there is no maximum or minimum score, score is D-score based on comparison of timing; positive scores equal more bias
Enhancing Assessment of Common Therapeutic factors | 6 months post-training
  Observed structured clinical evaluation using a standardized role play, minimum score = 0, maximum = 100, higher scores are better
Enhancing Assessment of Common Therapeutic factors | 3 months post-training
  Observed structured clinical evaluation using a standardized role play, minimum score = 0, maximum = 100, higher scores are better
Enhancing Assessment of Common Therapeutic factors | immediately after the training
  Observed structured clinical evaluation using a standardized role play, minimum score = 0, maximum = 100, higher scores are better
Social Distance Scale | 3 months post training
  12-item scale of willingness to interact with persons with mental illness, minimum = 0, maximum = 72, higher score is worse outcome
Social Distance Scale | immediately after the training
  12-item scale of willingness to interact with persons with mental illness, minimum = 0, maximum = 72, higher score is worse outcome
Patient: World Health Organization Disability Assessment Scale | 6-months post enrollment
  Assessment of daily functioning, minimum = 12, maximum = 60; higher score is worse
Patient: World Health Organization Disability Assessment Scale | 3-months post enrollment
  Assessment of daily functioning, minimum = 12, maximum = 60; higher score is worse
Patient Health Questionnaire 9 | 6-months post enrollment
  Depression symptoms, minimum = 0, maximum = 27, higher score is worse
Patient Health Questionnaire 9 | 3-months post enrollment
  Depression symptoms, minimum = 0, maximum = 27, higher score is worse
Patient: Generalized Anxiety Disorder 7 | 6 months post enrollment
  Anxiety symptoms, minimum = 0, maximum = 21, higher score is worse
Patient: Generalized Anxiety Disorder 7 | 3 months post enrollment
  Anxiety symptoms, minimum = 0, maximum = 21, higher score is worse
Patient: Positive and Negative Symptoms of Schizophrenia | 6 months post enrollment
  Psychosis symptoms, minimum = 0, maximum = 56, higher score is worse
Patient: Positive and Negative Symptoms of Schizophrenia | 3 months post enrollment
  Psychosis symptoms, minimum = 0, maximum = 56, higher score is worse
Patient: Alcohol Use Disorder Identification Test | 6-months post enrollment
  Alcohol Use Disorder symptoms, minimum = 0, maximum = 40, higher score is worse
Patient: Alcohol Use Disorder Identification Test | 3-months post enrollment
  Alcohol Use Disorder symptoms, minimum = 0, maximum = 40, higher score is worse
Patient: Euroqol 5 dimension 5 level | 6-months post enrollment
  Quality of life symptoms, minimum = 5, maximum=25, higher score is worse
Patient: Euroqol 5 dimension 5 level | 3-months post enrollment
  Quality of life symptoms, minimum = 5, maximum=25, higher score is worse
Patient: Cost of Service Receipt Inventory | 6-months post-enrollment
  Costs of care to patients, there is no maximum or minimum score, the outcome is total costs
Patient: Cost of Service Receipt Inventory | 3-months post-enrollment
  Costs of care to patients, , there is no maximum or minimum score, the outcome is total costs
Patient: Enhancing Assessment of Common Therapeutic factors | 6-months post-enrollment
  Common factors use by primary care provider, minimum score = 0, maximum = 15, higher score is better

CONTACTS AND LOCATIONS:
Overall Officials: Brandon A Kohrt, MD, PhD, Principal Investigator — George Washington University
Locations (1):
- Transcultural Psychosocial Organization Nepal, Pokhara, Gandaki, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Information will be shared through National Institute of Mental Health Data Archives
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available after publication of the primary and secondary outcomes manuscripts
Access Criteria: Managed through the National Institute of Mental Health Data Archives

REFERENCES:
- [Derived] Kohrt BA, Turner EL, Gurung D, Wang X, Neupane M, Luitel NP, Kartha MR, Poudyal A, Singh R, Rai S, Baral PP, McCutchan S, Gronholm PC, Hanlon C, Lempp H, Lund C, Thornicroft G, Gautam K, Jordans MJD. Implementation strategy in collaboration with people with lived experience of mental illness to reduce stigma among primary care providers in Nepal (RESHAPE): protocol for a type 3 hybrid implementation effectiveness cluster randomized controlled trial. Implement Sci. 2022 Jun 16;17(1):39. doi: 10.1186/s13012-022-01202-x. PMID 35710491